CLINICAL TRIAL: NCT05866250
Title: Dynamic Change of Doppler-based Renal Resistive Index in Predicting Renal Recovery From Acute Kidney Injury in Critically Ill Patients: a Prospective Observational Multicenter Study
Brief Title: Dynamic Change of Doppler-based Renal Resistive Index in Predicting Renal Recovery
Acronym: DRRRI
Status: Completed | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Dong Zhang, Director, The First Hospital of Jilin University
Other Study IDs: DongZhang
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; renal resistive index; prognosis; critically ill patients
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critically ill patients: All newly admitted ICU patients
  Interventions: Diagnostic Test: Doppler-based renal resistive index

INTERVENTIONS:
Diagnostic Test: Doppler-based renal resistive index — The kidney's interlobular or arcuate artery was preferentially selected and measured by pulse-wave Doppler.

SUMMARY:
The goal of this observational study is to observe the correlation between dynamic changes in the Doppler-based renal resistive index (RI) and the occurrence of persistent acute kidney injury (AKI) in critically ill patients. The main questions it aims to answer are:

* Are dynamic changes of RI within 24 or 48 hours associated with the prognosis of AKI (NO AKI, transient AKI, persistent AKI)?
* what are the influencing factors of changes in RI? Participants will measure values of RI in patients at admission (0 hour), after 24 hours and after 48 hours, respectively, and collect characters such as age, sex, vital signs, Apache II, diagnosis, renal function, applied drugs, fluid, 72-hour renal function and renal replacement, followed renal replacement and the mortality rate at 28 days.

DETAILED DESCRIPTION:
NO AKI is defined as No AKI occurred within 72 hour after ICU admission; Transient AKI is defined as AKI with recovery, which refers to the reduction in AKI stage ( (i.e., a decrease of serum creatinine, reversal of oliguria without diuretic therapy, and without need for renal replacement therapy) occurring with 72 hour after ICU admission; Persistent AKI is defined as AKI without recovery occurring with 72 hour after ICU admission.

ELIGIBILITY:
Inclusion Criteria:

• Patients admitted to the ICU within 24 h of admission.

Exclusion Criteria:

* Chronic kidney disease stage III-V;
* History of kidney transplantation;
* Previously known renal artery stenosis or renal vein thrombosis；
* Cardiac arrhythmia precluding renal Doppler measurement;
* Expected hospital stay < 72 h；
* Pregnant patients
* Last, patients with hospital stays < 72 h, since they could not be classified as having transient or persistent AKI according to our definitions, were secondarily excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the critically ill patients
Sampling Method: Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The prognosis of AKI | 72 hours
  NO AKI, transient AKI, persistent AKI. Transient AKI refers to the reduction in AKI stage ( (a decrease of serum creatinine, reversal of oliguria without diuretic therapy, and without need for renal replacement therapy) occurring with 72 hour after ICU admission. Persistent AKI refers to AKI without recovery occurring within 72 hours after ICU admission.

SECONDARY OUTCOMES:
Recovery of kidney function | 28 days
  A decrease of serum creatinine, reversal of oliguria without diuretic therapy, and without need for renal replacement therapy.
Mortality | 28 days
  Death or suivival

CONTACTS AND LOCATIONS:
Overall Officials: Dong Zhang, Director, Principal Investigator — The First Hospital of Jilin University
Locations (7):
- China (7):
  - Jilin Province People's Hospital, Changchun, Jlin
  - The First Hospital of Jilin University, Changchun, Jlin
  - The Third Affiliated Hospital of Changchung University, Changchun, Jlin
  - Dunhua City Hospital, Dunhua, Jlin
  - Jilin Central Hospital, Jilin, Jlin
  - Meihekou Central Hospital, Meihekou, Jlin
  - Jilin Siping Central People's Hospital, Siping, Jlin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Darmon M, Schortgen F, Vargas F, Liazydi A, Schlemmer B, Brun-Buisson C, Brochard L. Diagnostic accuracy of Doppler renal resistive index for reversibility of acute kidney injury in critically ill patients. Intensive Care Med. 2011 Jan;37(1):68-76. doi: 10.1007/s00134-010-2050-y. Epub 2010 Sep 23. PMID 20862450
- [Background] Saade A, Bourmaud A, Schnell D, Darmon M; R2D2 Study Group. Performance of Doppler-Based Resistive Index and Semiquantitative Renal Perfusion in Predicting Persistent Acute Kidney Injury According to Operator Experience: Post Hoc Analysis of a Prospective Multicenter Study. Crit Care Med. 2022 Apr 1;50(4):e361-e369. doi: 10.1097/CCM.0000000000005372. PMID 34678845
- [Background] Schnell D, Bourmaud A, Reynaud M, Rouleau S, Merdji H, Boivin A, Benyamina M, Vincent F, Lautrette A, Leroy C, Cohen Y, Legrand M, Morel J, Terreaux J, Darmon M. Performance of renal Doppler to predict the occurrence of acute kidney injury in patients without acute kidney injury at admission. J Crit Care. 2022 Jun;69:153983. doi: 10.1016/j.jcrc.2021.12.017. Epub 2022 Jan 21. PMID 35074631
- [Background] Darmon M, Bourmaud A, Reynaud M, Rouleau S, Meziani F, Boivin A, Benyamina M, Vincent F, Lautrette A, Leroy C, Cohen Y, Legrand M, Morel J, Terreaux J, Schnell D. Performance of Doppler-based resistive index and semi-quantitative renal perfusion in predicting persistent AKI: results of a prospective multicenter study. Intensive Care Med. 2018 Nov;44(11):1904-1913. doi: 10.1007/s00134-018-5386-3. Epub 2018 Oct 5. PMID 30291377